CLINICAL TRIAL: NCT02089165
Title: Randomized, Single-center, Open-label, Blinded Endpoint Assessment Study (Cross-over Study With 3 Study Products) on Bioavailability of Fatty Acids (Plasma Lipid Fractions) From Krill Oil and Krill Meal and Fatty Acids From Fish Oil in Healthy Subjects.
Brief Title: Bioavailability of Fatty Acids From Krill Oil and Krill Meal and Fatty Acids From Fish Oil in Healthy Subjects.
Acronym: RISU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Olympic Seafood AS (Industry)
Collaborators: Oy Foodfiles Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RISU 58/2013
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Krill oil (Experimental): The interventions are administered in the randomized order.
  Interventions: Dietary Supplement: Krill oil
- Krill meal (Experimental): The interventions are administered in the randomized order.
  Interventions: Dietary Supplement: Krill meal
- Fish oil (Active Comparator): The interventions are administered in the randomized order.
  Interventions: Dietary Supplement: Fish oil

INTERVENTIONS:
Dietary Supplement: Krill oil — Krill oil from Antarctic krill, per oral, capsule, targeted daily n-3 PUFA dose of 1 700 mg, single administration
  Arms: Krill oil
Dietary Supplement: Krill meal — Krill meal, granular meal from Antarctic krill, per oral, targeted daily n-3 PUFA dose of 1 700 mg, single administration
  Arms: Krill meal
Dietary Supplement: Fish oil — Fish oil, per oral, capsule, targeted daily n-3 PUFA dose of 1 700 mg, single administration
  Arms: Fish oil

SUMMARY:
The purpose of the study is to compare the acute bioavailability of two different krill oil products called krill oil and krill meal in comparison to fish oil product.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male
* Age 18 - 65 years
* Body mass index 18.5 - 30
* Informed consent, signed

Exclusion Criteria:

* Medication potential to affect the bioavailability of fatty acids (e.g. lipid-lowering drugs)
* Familial hypercholesterolemia, marked combined hyperlipidemia, condition that would impair, fat absorption (e.g. chronic pancreatitis, pancreatic lipase deficiency syndrome)
* Any untreated medical condition affecting absorption of fat
* Type 1 and 2 diabetes
* Cancer or other malignant disease within past five years
* Periodical hormone replacement therapy
* High intake of oily fish (once a week or more) (i.e. salmon, herring, sardines, mackerel, vendace)
* Smoking
* Alcohol consumption > 15 doses per week
* Females who are pregnant, breast-feeding or intend to become pregnant
* Hypersensitivity to any of the components of the test product
* Regular use of n-3 supplements 4 weeks before randomization
* Lack of suitability for participation in the trial, for any medical reason, as judged by the principal investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Incremental 0-72 h area under the curve of EPA + DHA proportion in plasma phospholipids. | 0-72 h

SECONDARY OUTCOMES:
Incremental 0-72 h area under the curve of EPA + DHA proportion in plasma triglyceride. | 0-72 h

OTHER OUTCOMES:
Mean proportions of fatty acids in plasma phospholipids and triglycerides. | 0-72 h

CONTACTS AND LOCATIONS:
Overall Officials: Essi S Sarkkinen, Ph.D, Study Director — Oy Foodfiles Ltd, member of Foodfiles group; Sakari A Nieminen, MD, Principal Investigator — Oy Foodfiles Ltd, memeber of Foodfiles group
Locations (1):
- Oy Foodfiles Ltd, memeber of Foodfiles group, Kuopio, Finland

REFERENCES:
- [Derived] Kohler A, Sarkkinen E, Tapola N, Niskanen T, Bruheim I. Bioavailability of fatty acids from krill oil, krill meal and fish oil in healthy subjects--a randomized, single-dose, cross-over trial. Lipids Health Dis. 2015 Mar 15;14:19. doi: 10.1186/s12944-015-0015-4. PMID 25884846